CLINICAL TRIAL: NCT06833099
Title: The Prediction of Recurrence Lumbar Disc Herniation At L5-S1 Level Through Machine Learning Models Based on Endoscopic Discectomy Via the Interlaminar Approach
Status: Completed | Type: Observational
Sponsor: Jinyu Chen (Other)
Collaborators: Nantong First People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Jinyu Chen, resident physician, Nantong First People's Hospital
Organization: Nantong First People's Hospital (Other)
Other Study IDs: JiajiaChen
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Lumbar Disc Herniation
Keywords: Machine Learning, Ensemble Learning
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biospecimen Description
  This study is a retrospective analysis that primarily uses clinical data and preoperative imaging records. Therefore, no biospecimens, such as blood or tissue samples, are collected, retained, or analyzed in this study. All data will be handled in strict accordance with privacy protection regulations set by the hospital's ethics committee and will be used exclusively by the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Recurrent rLDH: : Patients who experienced recurrent lumbar disc herniation following L5-S1 PEID.
  Interventions: Diagnostic Test: VAS Point and Imaging Examination
- Non-Recurrent rLDH: Patients who did not experience recurrent lumbar disc herniation following L5-S1 PEID.
  Interventions: Diagnostic Test: VAS Point and Imaging Examination

INTERVENTIONS:
Diagnostic Test: VAS Point and Imaging Examination — This intervention uses a machine learning model to predict the risk of recurrent lumbar disc herniation (rLDH) in patients who have had percutaneous endoscopic interlaminar discectomy (PEID) at the L5-S1 level. The model combines clinical data (e.g., BMI, disease duration, diabetes) and imaging metrics (e.g., posterior disc height index, spinal canal stenosis) to create a personalized risk score, unlike traditional methods that rely on clinical judgment or imaging alone.
  Key Features:
  Data-Driven Approach: Developed using data from 309 patients for real-world relevance.
  Advanced Variable Selection: Identifies eight key predictors using LASSO regression.
  Multiple Machine Learning Techniques: Uses algorithms like support vector machine, random forest, and extreme gradient boosting.
  Optimized for Clinical Decision-Making: Assists surgeons in personalizing treatment plans to reduce recurrence risk.

SUMMARY:
What Was the Study About? This study focused on improving the care of patients with a specific type of back problem called lumbar disc herniation at the L5-S1 level. Doctors often treat this condition with a minimally invasive surgery known as percutaneous endoscopic interlaminar discectomy (PEID). However, sometimes the herniation (the damaged disc) can come back after surgery. The goal of this study was to develop computer models that help predict which patients might experience a recurrence of their herniated disc.

Who Participated? The study reviewed the medical records of 309 patients who had undergone the PEID surgery. Out of these, 33 patients experienced a recurrence of their herniation, while 276 patients did not.

What Did the Researchers Do?

Data Collection:

They gathered information from each patient before the surgery, including clinical details (like body weight and any health conditions such as diabetes) and imaging studies (like X-rays, CT scans, or MRIs) that show the condition of the spine.

Identifying Key Risk Factors:

Using a statistical method called LASSO regression, the researchers identified eight important factors that could influence whether the herniation might come back. These included factors such as body mass index (BMI), a measure related to disc height (posterior disc height index), signs of spinal canal narrowing, how long the patient had symptoms before surgery, and other health conditions.

Developing Prediction Models:

They then used several machine learning techniques (advanced computer methods that learn from data) to build prediction models. Two of the best-performing models were based on methods called Random Forest and Extreme Gradient Boosting (XGB).

What Were the Main Findings?

Key Predictors: Higher BMI and changes in the disc (as measured by the posterior disc height index) were found to be the strongest predictors of a herniation coming back after surgery. Other factors, like spinal canal narrowing and longer duration of symptoms before surgery, also played significant roles.

Practical Implication: These models can help doctors identify which patients are at higher risk for recurrence. With this information, they can adjust treatment plans and follow-up care to better manage and potentially reduce the risk of the herniation coming back.

Why Is This Important? For patients and their families, this study offers hope for more personalized and effective treatment plans, reducing the chances of needing additional surgeries in the future. For healthcare providers, the findings provide useful tools to improve decision-making before surgery, ensuring better long-term outcomes for patients with L5-S1 lumbar disc herniation.

In summary, this research uses modern computer methods to predict the risk of recurrent disc herniation after a common minimally invasive back surgery, aiming to enhance patient care and improve surgical outcomes.

DETAILED DESCRIPTION:
Detailed Description

This study aimed to enhance care for patients undergoing a minimally invasive spine surgery known as percutaneous endoscopic interlaminar discectomy (PEID), which is used to treat herniated discs at the L5-S1 level. Recurrent disc herniation-where the disc problem returns after surgery-can lead to additional pain and the need for further treatment. To address this issue, the research team conducted an in-depth review of patient data gathered at a single hospital.

How the Study Was Conducted Researchers collected comprehensive information from 309 patients who had undergone PEID. This information included clinical details (such as age, body mass index, and existing conditions like diabetes) and imaging data (from X-rays, CT scans, and MRIs) that provided insights into the structure and condition of the spine. Rather than relying on a single factor, the study examined a wide range of variables to understand which ones might predict a recurrence of the herniated disc.

Advanced Data Analysis and Prediction Methods To sift through the large amount of collected data, the team used a statistical technique called LASSO regression. This method helped identify the most influential factors from many possible measurements. Eight key factors emerged, including body mass index (BMI) and specific measurements related to the spinal disc's structure.

Building on this foundation, the study employed several machine learning techniques-advanced computer methods that detect patterns in data-to create models capable of predicting the risk of recurrence. Among the various models tested, two (Random Forest and Extreme Gradient Boosting) stood out for their strong performance. These models not only highlighted the significance of factors like BMI and certain spinal measurements but also provided a promising tool for clinicians to assess risk before surgery.

Why This Matters For healthcare providers, having a reliable predictive model means they can better tailor surgical techniques and postoperative care to individual patients. By understanding a patient's risk profile, surgeons can take additional precautions or consider alternative approaches to reduce the chance of recurrence. For patients and their families, this translates into more personalized treatment plans and potentially fewer complications or repeat surgeries in the future.

In Summary This study represents an important step toward personalized medicine in spinal care. By integrating detailed clinical and imaging data with state-of-the-art machine learning techniques, the researchers developed a model that can forecast the likelihood of a recurrent herniated disc after PEID surgery. The insights gained not only improve the understanding of key risk factors but also pave the way for more targeted and effective treatment strategies, ultimately aiming to enhance long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for rLDH: (A) Patients with L5-S1 lumbar disc herniation who underwent single level PEID. (B) Completed comprehensive imaging examinations within one month before surgery.

(C) Postoperative VAS scores decreased by ≥60%, followed by an increase, confirmed by imaging.

(D) No other abnormalities detected in imaging. (E) Minimum follow-up period of 6 months.

Inclusion Criteria for Non-rLDH: (A) Patients with L5-S1 lumbar disc herniation who underwent single-level PEID. (B) Completed comprehensive imaging examinations within one month before surgery. (C) Postoperative VAS scores decreased by ≥60% without recurrence. (D) No other abnormalities detected in imaging. (E) Minimum follow-up period of 6 months.

Exclusion Criteria:

(A) Presence of other pathological conditions causing lower back pain, such as disc infections, spinal tumors, metabolic bone disease, or osteoporosis. (B) History of prior lumbar disc or other spinal surgeries. (C) Poor imaging quality or incomplete examination data. (D) Patients lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population Description:
  The study population consisted of 309 patients who underwent percutaneous endoscopic interlaminar discectomy (PEID) for L5-S1 lumbar disc herniation between January 2020 and June 2024 at Nantong First People's Hospital. All patients had at least 6 months of follow-up post-surgery. The study focused on identifying factors that predict recurrent lumbar disc herniation (rLDH) after the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of Lumbar Disc Herniation (rLDH) Following Percutaneous Endoscopic Interlaminar Discectomy (PEID) at the L5-S1 Level | The recurrence will be monitored and documented during follow-up visits at least 6 months
  The primary outcome measure will assess the recurrence of lumbar disc herniation (rLDH) in patients who have undergone percutaneous endoscopic interlaminar discectomy (PEID) at the L5-S1 level. The occurrence of rLDH will be evaluated based on clinical symptoms and imaging findings, including MRI or CT scans, within a specified follow-up period post-surgery. This measure aims to develop a predictive model to estimate the likelihood of recurrence of disc herniation following PEID at the L5-S1 level.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantong First People's Hospital, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of patient clinical and imaging data, and to protect patient privacy and data security, we do not plan to share individual participant data (IPD) with other researchers. Sharing such data could potentially lead to the leakage of personal information, so we have decided not to make these data publicly available. All data will be handled in strict accordance with privacy protection regulations set by the hospital's ethics committee and will be used exclusively within the research team.

REFERENCES:
- [Background] Shi H, Zhu L, Jiang ZL, Wu XT. Radiological risk factors for recurrent lumbar disc herniation after percutaneous transforaminal endoscopic discectomy: a retrospective matched case-control study. Eur Spine J. 2021 Apr;30(4):886-892. doi: 10.1007/s00586-020-06674-3. Epub 2021 Jan 1. PMID 33386474
- [Background] Yu C, Zhan X, Liu C, Liao S, Xu J, Liang T, Zhang Z, Chen J. Risk Factors for Recurrent L5-S1 Disc Herniation After Percutaneous Endoscopic Transforaminal Discectomy: A Retrospective Study. Med Sci Monit. 2020 Mar 25;26:e919888. doi: 10.12659/MSM.919888. PMID 32210223
- [Background] Choi G, Lee SH, Raiturker PP, Lee S, Chae YS. Percutaneous endoscopic interlaminar discectomy for intracanalicular disc herniations at L5-S1 using a rigid working channel endoscope. Neurosurgery. 2006 Feb;58(1 Suppl):ONS59-68; discussion ONS59-68. doi: 10.1227/01.neu.0000192713.95921.4a. PMID 16479630
- [Background] Siemionow K, An H, Masuda K, Andersson G, Cs-Szabo G. The effects of age, sex, ethnicity, and spinal level on the rate of intervertebral disc degeneration: a review of 1712 intervertebral discs. Spine (Phila Pa 1976). 2011 Aug 1;36(17):1333-9. doi: 10.1097/BRS.0b013e3181f2a177. PMID 21217432
- [Background] Li Y, Wang B, Li H, Chang X, Wu Y, Hu Z, Liu C, Gao X, Zhang Y, Liu H, Li Y, Li C. Adjuvant surgical decision-making system for lumbar intervertebral disc herniation after percutaneous endoscopic lumber discectomy: a retrospective nonlinear multiple logistic regression prediction model based on a large sample. Spine J. 2021 Dec;21(12):2035-2048. doi: 10.1016/j.spinee.2021.07.012. Epub 2021 Jul 20. PMID 34298160
- [Background] Jia M, Sheng Y, Chen G, Zhang W, Lin J, Lu S, Li F, Ying J, Teng H. Development and validation of a nomogram predicting the risk of recurrent lumbar disk herniation within 6 months after percutaneous endoscopic lumbar discectomy. J Orthop Surg Res. 2021 Apr 21;16(1):274. doi: 10.1186/s13018-021-02425-2. PMID 33882995
- [Background] Han M, Liu L, Hu M, Liu G, Li P. Medical expert and machine learning analysis of lumbar disc herniation based on magnetic resonance imaging. Comput Methods Programs Biomed. 2022 Jan;213:106498. doi: 10.1016/j.cmpb.2021.106498. Epub 2021 Oct 29. PMID 34758430
- [Background] Li R, Fu D, Han H, Zhan Z, Wu Y, Meng B. Comparative analysis of percutaneous endoscopic interlaminar discectomy for highly downward-migrated disc herniation. J Orthop Surg Res. 2023 Aug 14;18(1):602. doi: 10.1186/s13018-023-04090-z. PMID 37580753
- [Background] Berg B, Gorosito MA, Fjeld O, Haugerud H, Storheim K, Solberg TK, Grotle M. Machine Learning Models for Predicting Disability and Pain Following Lumbar Disc Herniation Surgery. JAMA Netw Open. 2024 Feb 5;7(2):e2355024. doi: 10.1001/jamanetworkopen.2023.55024. PMID 38324310
- [Background] Harada GK, Siyaji ZK, Mallow GM, Hornung AL, Hassan F, Basques BA, Mohammed HA, Sayari AJ, Samartzis D, An HS. Artificial intelligence predicts disk re-herniation following lumbar microdiscectomy: development of the "RAD" risk profile. Eur Spine J. 2021 Aug;30(8):2167-2175. doi: 10.1007/s00586-021-06866-5. Epub 2021 Jun 7. PMID 34100112
- [Background] Wang H, Zhou Y, Li C, Liu J, Xiang L. Risk factors for failure of single-level percutaneous endoscopic lumbar discectomy. J Neurosurg Spine. 2015 Sep;23(3):320-5. doi: 10.3171/2014.10.SPINE1442. Epub 2015 Jun 12. PMID 26068272
- [Background] Huang W, Han Z, Liu J, Yu L, Yu X. Risk Factors for Recurrent Lumbar Disc Herniation: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2016 Jan;95(2):e2378. doi: 10.1097/MD.0000000000002378. PMID 26765413
- [Background] Li H, Deng W, Wei F, Zhang L, Chen F. Factors related to the postoperative recurrence of lumbar disc herniation treated by percutaneous transforaminal endoscopy: A meta-analysis. Front Surg. 2023 Jan 19;9:1049779. doi: 10.3389/fsurg.2022.1049779. eCollection 2022. PMID 36743903
- [Background] Ren G, Liu L, Zhang P, Xie Z, Wang P, Zhang W, Wang H, Shen M, Deng L, Tao Y, Li X, Wang J, Wang Y, Wu X. Machine Learning Predicts Recurrent Lumbar Disc Herniation Following Percutaneous Endoscopic Lumbar Discectomy. Global Spine J. 2024 Jan;14(1):146-152. doi: 10.1177/21925682221097650. Epub 2022 May 2. PMID 35499394
- [Background] Modic MT, Ross JS. Lumbar degenerative disk disease. Radiology. 2007 Oct;245(1):43-61. doi: 10.1148/radiol.2451051706. PMID 17885180
- [Background] Ju CI, Lee SM. Complications and Management of Endoscopic Spinal Surgery. Neurospine. 2023 Mar;20(1):56-77. doi: 10.14245/ns.2346226.113. Epub 2023 Mar 31. PMID 37016854
- [Background] Pan M, Li Q, Li S, Mao H, Meng B, Zhou F, Yang H. Percutaneous Endoscopic Lumbar Discectomy: Indications and Complications. Pain Physician. 2020 Jan;23(1):49-56. PMID 32013278
- [Background] Yin S, Du H, Yang W, Duan C, Feng C, Tao H. Prevalence of Recurrent Herniation Following Percutaneous Endoscopic Lumbar Discectomy: A Meta-Analysis. Pain Physician. 2018 Jul;21(4):337-350. PMID 30045591
- [Background] Cheng J, Wang H, Zheng W, Li C, Wang J, Zhang Z, Huang B, Zhou Y. Reoperation after lumbar disc surgery in two hundred and seven patients. Int Orthop. 2013 Aug;37(8):1511-7. doi: 10.1007/s00264-013-1925-2. Epub 2013 May 22. PMID 23695881
- [Background] Chen Z, Wang X, Cui X, Zhang G, Xu J, Lian X. Transforaminal Versus Interlaminar Approach of Full-Endoscopic Lumbar Discectomy Under Local Anesthesia for L5/S1 Disc Herniation: A Randomized Controlled Trial. Pain Physician. 2022 Nov;25(8):E1191-E1198. PMID 36375189